CLINICAL TRIAL: NCT02496884
Title: A Randomized, Double-blind, Placebo-controlled Safety Study of DS-5565 for Treatment of Pain Due to Fibromyalgia in Subjects With Chronic Kidney Disease
Brief Title: Safety Study of DS-5565 for Treatment of Fibromyalgia Pain in Subjects With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS5565-A-U307; 2014-003972-21 (EudraCT Number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Fibromyalgia
Keywords: chronic kidney disease; . α2δ ligands; mirogabalin; pain relief; kidney metabolism
MeSH Terms: conditions — Fibromyalgia; Renal Insufficiency, Chronic | interventions — mirogabalin; Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- M-CKD DS-5565 7.5 mg BID (Experimental): Patients with moderate chronic kidney disease (M-CKD) randomized to receive DS-5565 BID during the treatment period.
  Interventions: Drug: DS-5565
- S-CKD DS-5565 7.5 mg QD (Experimental): Fibromyalgia patients with severe chronic kidney disease (S-CKD) randomized to receive a DS-5565 7.5 mg tablet once per day (QD), and a placebo tablet (no drug) QD, for a total of 7.5 mg DS-5565
  Interventions: Drug: DS-5565; Drug: Placebo
- M-CKD Placebo (Placebo Comparator): Patients with M-CKD randomized to receive placebo twice daily (BID) during the treatment period.
  Interventions: Drug: Placebo
- S-CKD Placebo (Placebo Comparator): Patients with S-CKD randomized to receive placebo once daily (QD) during the treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-5565 — DS-5565 7.5 mg tablet for oral use
  Other Names: Experimental drug; Mirogabalin; SUB60040
  Arms: M-CKD DS-5565 7.5 mg BID; S-CKD DS-5565 7.5 mg QD
Drug: Placebo — Placebo tablet for oral use to match DS-5565 7.5 mg tablet
  Other Names: No drug; Placebo comparator
  Arms: M-CKD Placebo; S-CKD DS-5565 7.5 mg QD; S-CKD Placebo

SUMMARY:
DS-5565 (mirogabalin) is being studied as treatment for fibromyalgia (FM) pain. Because it is excreted through the kidneys, people who have reduced kidney function will not process the drug as well as with those with normal kidney function, so the dose must be reduced. This study will test two reduced dose levels for both moderately reduced and severely reduced kidney function. The study will test the hypothesis that the drug will be safe and well-tolerated in people who have both fibromyalgia and chronic kidney disease.

DETAILED DESCRIPTION:
The main objective of the trial is to determine the safety and tolerability of subjects with FM and moderate to severe renal dysfunction during 13 weeks of renally-adjusted dosing of DS-5565 compared to placebo, followed by a short-term (4-week) safety follow-up.

This trial is conducted in accordance with the ethical principles of Good Clinical Practice, according to the International Council for Harmonisation (ICH) Harmonised Tripartite Guidelines. An independent Data Safety Monitoring Board (DSMB) is created to further protect the rights, safety, and well-being of subjects who participate in this study by monitoring their progress and results. The independent DSMB is composed of qualified scientists who are not investigators in the study and not otherwise directly associated with the sponsor.

Additional protection is provided by special monitoring of liver enzyme elevations and liver dysfunction performed by a Hepatic Adjudication Committee (HAC), comprised of three qualified hepatologists who are not investigators in the study and not otherwise directly associated with the sponsor. The HAC completes assessments on an ongoing basis. Adjudication of hepatic events is based on evaluation of electronic case report forms (eCRFs) and source documents, as available, including but not limited to hospital discharge summaries, diagnostic imaging, histopathology, consultation, and laboratory reports.

ELIGIBILITY:
Abbreviations: alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine clearance [(CrCL) determined by the central laboratory using the Cockcroft-Gault equation], upper limit of normal (ULN), Columbia-Suicide Severity Rating Scale (C-SSRS)

Inclusion Criteria:

* Age ≥ 18 years
* Able to give written informed consent
* Able to complete patient-reported questionnaires per the Investigator's judgment
* Estimated CrCl between 15-59 mL/min from serum creatinine by the central laboratory using the Cockcroft-Gault equation
* Fibromyalgia meeting American College of Rheumatology criteria for FM:

  * Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5 or WPI 3 to 6 and SS scale score ≥ 9,
  * Pain in at least 11 of 18 specific tender point sites,
  * Symptoms have been present at a similar level for at least 3 months, and
  * The subject does not have a disorder that would otherwise explain the pain
* Average Daily Pain Score of ≥ 4 on the 11-point numeric rating scale (NRS) over the 7 days prior to randomization (based on completion of at least 4 daily pain assessments during the 7-day baseline period prior to randomization)
* Women of child bearing potential (WOCBP) must be using adequate methods of contraception to avoid pregnancy during the study and for 4 weeks after study completion.

Exclusion Criteria:

* Need for ongoing use of concomitant chronic pain medications or any new non-pharmacological pain management techniques that may confound assessments of efficacy and/or safety, including neurolytic treatments (destruction of nerves by chemicals, heat, cold) or surgery, intrathecal pumps, spinal cord stimulators or psychological support within the previous year. Also excluded: topical capsaicin within 6 months; or systemic corticosteroids within 3 months of baseline period.
* Unable to undergo pre-study washout of prohibited concomitant medications
* Subjects with recent history (i.e., within 1 year prior to screening) of alcohol abuse or illicit drug use (cocaine, heroin, marijuana [including medical, prescribed], etc.)
* Use of any selective serotonin reuptake inhibitor (SSRI), unless the subject has been on a stable dose for ≥ 90 days prior to screening and is not anticipated to need any dose adjustment during the course of the study
* Subjects with severe or uncontrolled depression that, in the judgment of the Investigator, makes the subject inappropriate for entry into the study
* Significant neurological or psychiatric disorder unrelated to neuropathic pain
* Other severe pain (eg, sciatica, rheumatoid arthritis) that might impair the assessment of neuropathic pain
* CrCl ≥ 60 mL/min estimated from serum creatinine by the central laboratory using the Cockcroft-Gault equation.
* Subjects who are on hemodialysis or who require hemodialysis before the follow-up assessment; acute renal failure; history of kidney transplant
* Any history of a malignancy other than basal cell carcinoma within the past 5 years
* Clinically significant unstable neurologic, ophthalmologic, hepatobiliary, respiratory, or hematologic illness or unstable cardiovascular disease (eg, severe hypotension, uncontrolled cardiac arrhythmia, or myocardial infarction) within 12 months prior to screening
* Pregnancy or breast feeding or intent to become pregnant during the study period
* Known hypersensitivity to α2δ ligands or other components of the study medications. Note: Prior exposure to DS-5565 is allowed, as long as hypersensitivity to DS-5565 was not observed.
* Clinically significant ECG abnormalities at the Screening Visit
* Subjects who are at risk of suicide, as defined by their responses to the C-SSRS or in the opinion of the Investigator. Note: Subjects answering "yes" to any of the questions about active suicidal ideation/intent/behaviors that occurred within the past 12 months must be excluded (C-SSRS Suicide Ideation section - Questions 3, 4, or 5; C-SSRS Suicidal Behavior section - any of the suicide behaviors questions). Such subjects should be referred immediately to a mental health professional for appropriate evaluation.
* Subjects who are unlikely to comply with the protocol (eg, uncooperative attitude, inability to return for subsequent visits, and/or otherwise considered by the Investigator to be unlikely to complete the study)
* Subject is currently enrolled in, or it has been fewer than 30 days since ending, another investigational device or drug study or is receiving another investigational agent.
* Subjects who are employees or immediate family of employees of the study site, Sponsor, or contract research organization (CRO)
* Screening laboratory values outside the limits listed in the table below:

  * Hematology
  * Hemoglobin < 8 g/dL
  * Platelet count < 100,000/mm3
  * Absolute neutrophil count < 1,500/mm3
  * Blood chemistry
  * AST > 2.0 × ULN
  * ALT > 2.0 × ULN
  * Alkaline phosphatase > 1.5 × ULN
  * Total bilirubin > 1.2 × ULN (If a subject has total bilirubin >ULN: unconjugated and conjugated bilirubin fractions should be analyzed and only subject documented to have Gilbert's syndrome may be enrolled)
  * Creatine kinase > 3.0 × ULN
  * Calculated CrCl ≥ 60 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (39):
- United States (22):
  - Phoenix, Arizona
  - Colton, California
  - Los Angeles, California
  - Santa Ana, California
  - Colorado Springs, Colorado
  - Brooksville, Florida
  - DeBary, Florida
  - Hialeah, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Grand Blanc, Michigan
  - High Point, North Carolina
  - Cincinnati, Ohio
  - Wyomissing, Pennsylvania
  - Greer, South Carolina
  - Rapid City, South Dakota
  - Knoxville, Tennessee
  - Houston, Texas
  - Plano, Texas
  - Bellevue, Washington
  - Charleston, West Virginia
  - Morgantown, West Virginia
- Bulgaria (5):
  - Plovdiv
  - Sevlievo
  - Sofia
  - Stara Zagora
  - Varna
- Czechia (2):
  - Prague
  - Říčany
- Hungary (2):
  - Budapest
  - Nyíregyháza
- Poland (2):
  - Elblag
  - Krakow
- Cluj-Napoca, Romania
- South Africa (2):
  - Johannesburg
  - Pretoria
- Spain (3):
  - Barcelona
  - Santiago de Compostela
  - Valencia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 participants who met all inclusion and no exclusion criteria were randomized to treatment in four countries: Bulgaria, Romania, Spain, and the United States.
Pre-assignment Details: Eligible participants were randomized 2:1 to receive either DS-5565 7.5 mg QD or placebo for participants with CrCl 15 to 29 mL/min, or 2:1 to receive treatment with DS-5565 7.5 mg BID or placebo for participants with CrCl 30 to 59 mL/min over a 13-week double-blind treatment period.
Groups:
- M-CKD Placebo: Patients with moderate chronic kidney disease (M-CKD) randomized to receive placebo twice daily (BID) during the treatment period.
- M-CKD DS-5565 7.5 mg BID: Patients with moderate chronic kidney disease (M-CKD) randomized to receive DS-5565 7.5 mg BID during the treatment period.
- S-CKD Placebo: Patients with severe chronic kidney disease (S-CKD) randomized to receive placebo once daily (QD) during the treatment period.
- S-CKD DS-5565 7.5 mg QD: Patients with severe chronic kidney disease (S-CKD) randomized to receive a DS-5565 7.5 mg tablet once per day (QD).
Period: Overall Study
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD
Started | 17 | 34 | 1 | 4
Safety Analysis Set | 17 | 34 | 1 | 4
Modified Intent to Treat Set (mITT) | 17 | 34 | 1 | 4
Pharmacokinetic (PK) Analysis Set | 0 | 33 | 0 | 4
Completed Treatment Per Protocol | 16 | 27 | 1 | 3
Completed | 15 | 31 | 1 | 4
Not Completed | 2 | 3 | 0 | 0
Not completed — Counted twice as enrolled | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics are reported in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD | Total
Number analyzed (Participants) | 17 | 34 | 1 | 4 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 1 | 1 | 22
  >=65 years | 9 | 22 | 0 | 3 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.39) | 68.4 (13.92) | 53.0 | 74.0 (12.25) | 67.3 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 28 | 1 | 0 | 45
  Male | 1 | 6 | 0 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 1 | 6
  White | 14 | 29 | 0 | 2 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Average Daily Pain Score (ADPS) [Count of Participants; unit: Participants] — Participants were asked to rate their pain on a scale of 0-10, where 0=no pain and 10=the most pain experienced. The average ADPS at baseline was recorded.
  Participants
    ADPS less than 7 | 8 | 9 | 1 | 2 | 20
    ADPS 7 or more | 9 | 25 | 0 | 2 | 36
Baseline Average Daily Pain Score (ADPS) [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to rate their pain on a scale of 0-10, where 0=no pain and 10=the most pain experienced, where higher scores indicate worse outcome. The average ADPS at baseline was recorded.
  units on a scale | 6.99 (1.35) | 7.21 (0.96) | 5.70 | 6.53 (0.82) | 7.07 (1.09)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Treatment Emergent Adverse Event (TEAE)
Description: A TEAE is any adverse event that emerges on or after the first dosing of double blind study medication and during study treatment up to 4 weeks after the last dose of double blind study medication (having been absent prior to treatment) or worsens relative to the pre-double blind treatment state. Relationship of TEAEs to study drug is assessed by the investigator.
  Clinically significant changes from baseline in clinical laboratory evaluations, neurological examinations, and electrocardiograms are reported as TEAEs.
Time Frame: Baseline up to 30 days after last dose, up to 25 months
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD
Number analyzed (Participants) | 17 | 34 | 1 | 4
Participants
  At least 1 TEAE | 8 | 16 | 0 | 3
  Drug-related TEAEs | 1 | 9 | 0 | 0
  Serious TEAE | 0 | 1 | 0 | 0
  Drug-related serious TEAE | 0 | 0 | 0 | 0

2. Primary Outcome: Patients Answering Yes to Any Question on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is described as a scale developed at Columbia University that has 2-6 questions each in categories of Suicidal Ideation, Intensity of Ideation, Suicidal Behavior, and Actual Attempts. Four constructs were measured. Severity of Suicidal ideation is rated on a 5-point ordinal scale. Intensity of ideation is comprised of 5 items (frequency, duration, controllability, deterrents, and reason for ideation), each rated on a 5-point ordinal scale. Suicidal behavior is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal self-injurious behavior. Lethality, assesses actual attempts; actual lethality is rated on a 6-point ordinal scale, and if actual lethality is 0, potential lethality of attempts is rated on a 3-point ordinal scale.The higher the C-SSRS score, the higher the suicide risk (ie. worse outcome).
Time Frame: Screening up to Week 13 postdose
Population: The C-SSRS score was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD
Number analyzed (Participants) | 17 | 34 | 1 | 4
Participants
  Screening | 0 | 0 | 0 | 0
  Baseline | 0 | 0 | 0 | 0
  Week 13 | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Weekly Average of Individual Daily Pain Scores (ADPS)
Description: Each day participants will rate their worst pain over the last 24 hours on a scale from 0-10, where 0=no pain and 10=worst pain imaginable. Each week individual pain scores will be averaged, and the mean weekly score for the treatment group will be calculated. Higher ADPS scores indicate worse outcome.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11, Week 12, and Week 13 postdose
Population: Average daily pain scores were assessed in the modified Intent-to-Treat (mITT) Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD
Number analyzed (Participants) | 17 | 34 | 1 | 4
units on a scale
  Baseline | 6.99 (1.35) | 7.21 (0.96) | 5.70 | 6.53 (0.82)
  Week 1 | 6.26 (1.53) | 6.10 (1.63) | 2.0 | 6.88 (0.15)
  Week 2 | 6.03 (1.68) | 5.73 (2.06) | 1.70 | 6.60 (0.80)
  Week 3 | 5.77 (1.72) | 5.55 (1.94) | 1.70 | 6.80 (0.40)
  Week 4 | 5.41 (1.91) | 5.43 (1.99) | 1.30 | 6.75 (0.50)
  Week 5 | 5.45 (1.65) | 5.46 (2.08) | 0.70 | 6.90 (0.99)
  Week 6 | 5.16 (1.75) | 5.16 (2.18) | 1.4 | 6.43 (1.91)
  Week 7 | 5.03 (2.10) | 5.09 (2.14) | 1.20 | 6.67 (1.53)
  Week 8 | 5.15 (2.03) | 5.04 (2.23) | 1.00 | 6.73 (1.52)
  Week 9 | 5.09 (1.82) | 4.81 (2.24) | 1.00 | 6.47 (1.91)
  Week 10 | 4.86 (2.06) | 4.97 (2.20) | 0.90 | 6.53 (1.75)
  Week 11 | 4.28 (1.99) | 4.80 (2.31) | 0.70 | 6.73 (1.12)
  Week 12 | 4.17 (2.16) | 4.69 (2.20) | 0.80 | 6.63 (2.27)
  Week 13 | 4.28 (2.45) | 4.15 (1.84) | 1.00 | 6.80 (2.23)

4. Secondary Outcome: Number of Participants With Different Scale Ranges of the Patient Global Impression of Change (PGIC) Scale at Week 13
Description: The PGIC is a validated outcome measure for treatment of pain in the acute pain setting. At the end of treatment, participants will rate their overall status on a scale of 1-7, where 1=very much improved and 7=very much worse using the standard PGIC questionnaire. Higher scores indicate worse outcome.
Time Frame: Week 13 postdose
Population: Patient Global Impression of Change (PGIC) scores were assessed in the modified Intent-to-Treat (mITT) Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD
Number analyzed (Participants) | 17 | 34 | 1 | 4
Participants
  Score 1-3; Improved | 12 | 20 | 1 | 1
  Score 4; No change | 3 | 8 | 0 | 3
  Score 5-7; Worsened | 1 | 0 | 0 | 0
  Missing | 1 | 6 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days after last dose, up to 25 months.
Description: A TEAE was any adverse event that emerged on or after the first dosing of double-blind study medication and during study treatment up to 4 weeks after the last dose of double-blind study medication (having been absent prior to treatment) or worsened relative to the pre-double-blind treatment state.
Arm/Group | M-CKD Placebo | M-CKD DS-5565 7.5 mg BID | S-CKD Placebo | S-CKD DS-5565 7.5 mg QD
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/34 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/34 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 8/17 | 16/34 | 0/1 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M-CKD Placebo (N=17) | M-CKD DS-5565 7.5 mg BID (N=34) | S-CKD Placebo (N=1) | S-CKD DS-5565 7.5 mg QD (N=4)
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M-CKD Placebo (N=17) | M-CKD DS-5565 7.5 mg BID (N=34) | S-CKD Placebo (N=1) | S-CKD DS-5565 7.5 mg QD (N=4)
Drug withdrawal syndrome (General disorders) | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 2 | 0 | 0
Creatinine renal decreased (Investigations) | 1 | 0 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT02496884/Prot_SAP_000.pdf